CLINICAL TRIAL: NCT02854046
Title: Calciphylaxis : Population, Risk Factors, Diagnostic Practice, Therapeutic and Outcome : a Multicentric, Retrospective Cohort
Brief Title: Calciphylaxis : Population, Risk Factors, Diagnostic Practice, Therapeutic and Outcome
Acronym: CalciWest
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0164
Record Dates: First submitted 2016-07-26; First posted 2016-08-03 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Calciphylaxis
Keywords: calcific uremic arteriolopathy; case-control study; cohort study
MeSH Terms: conditions — Calciphylaxis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Calciphylaxis Cases: Adult patients with advanced chronic kidney disease (DFG estimation < 30 ml/min/1.73m² - beyond 3B stage) with/without substitute therapy who has presented a case of calciphylaxis (Calcific Uremic Arteriolopathy) between 2006 and 2016 in the Regions of Pays de la Loire, Centre Val de Loire, Bretagne and Poitou-Charentes
  Interventions: Other: Calcific Uremic Arteriolopathy
- Witness cases: Selected anonymously in French national register REIN. Matched to Calciphylaxis Cases according to gender, age, treatment by extrarenal purification at the timepoint "onset of the lesions" and REIN regions belonging

INTERVENTIONS:
Other: Calcific Uremic Arteriolopathy
  Groups: Calciphylaxis Cases

SUMMARY:
Calciphylaxis, also called Calcific Uremic Arteriolopathy (CUA) is a lethal affection mostly affecting patient in end stage renal disease. The survival rate is described around 20 to 46% at one year.

Clinical presentation is very painful skin lesions with ulceration mostly located on the trunk or thigh.

Current knowledge about physiopathology, diagnostic practice and therapeutic is very limited.

Actually there is no European study about calciphylaxis and risk factors, diagnostic practice and outcome factors.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years with chronic renal failure with Glomerular Filtration Rate < 30ml/min/1,73m²
* diagnosis of calciphylaxis between 2006 and 2016
* living in the Regions of Bretagne, Pays de la Loire, Poitou-Charentes or Centre Val de Loire.

Exclusion Criteria:

* realized biopsy in favor of differential diagnosis
* significant arterial lesion of lesion area or differential diagnosis more valid
* if the diagnosis is not based on the following criteria: 3 clinical criteria or 2 clinical criteria and biopsy in favor, criteria which are :

  * Patient in chronic hemodialysis or stade 4 chronic kidney disease
  * At least 2 painful sores and hardly curable with concomitant painful purpura
  * Sore and purpura localisation in trunk, extremities and penis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced chronic kidney disease (DFG estimation < 30 ml/min/1.73m² - beyond 3B stage) with/without subtitute therapy who has presented a case of calciphylaxis between 2006 and 2016 in the Régions of Pays de la Loire, Centre Val de Loire, Bretagne and Poitou-Charentes
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Description of calcific uremic arteriolopathy in a French population by describing the characteristics of the population, diagnostic and treatment practices and patient outcome. | Up to 16 months

SECONDARY OUTCOMES:
Study factors determining the patient outcome with calciphylaxis | Up to 16 months
Study case control of risk factors in the subgroup of patients in extra renal replacement therapy | Up to 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryvonne HOURMANT, PHD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandenburg VM, Kramann R, Rothe H, Kaesler N, Korbiel J, Specht P, Schmitz S, Kruger T, Floege J, Ketteler M. Calcific uraemic arteriolopathy (calciphylaxis): data from a large nationwide registry. Nephrol Dial Transplant. 2017 Jan 1;32(1):126-132. doi: 10.1093/ndt/gfv438. PMID 26908770
- [Background] Floege J, Kubo Y, Floege A, Chertow GM, Parfrey PS. The Effect of Cinacalcet on Calcific Uremic Arteriolopathy Events in Patients Receiving Hemodialysis: The EVOLVE Trial. Clin J Am Soc Nephrol. 2015 May 7;10(5):800-7. doi: 10.2215/CJN.10221014. Epub 2015 Apr 17. PMID 25887067
- [Background] Fine A, Zacharias J. Calciphylaxis is usually non-ulcerating: risk factors, outcome and therapy. Kidney Int. 2002 Jun;61(6):2210-7. doi: 10.1046/j.1523-1755.2002.00375.x. PMID 12028462
- [Background] Weenig RH, Sewell LD, Davis MD, McCarthy JT, Pittelkow MR. Calciphylaxis: natural history, risk factor analysis, and outcome. J Am Acad Dermatol. 2007 Apr;56(4):569-79. doi: 10.1016/j.jaad.2006.08.065. Epub 2006 Dec 1. PMID 17141359
- [Derived] Gaisne R, Pere M, Menoyo V, Hourmant M, Larmet-Burgeot D. Calciphylaxis epidemiology, risk factors, treatment and survival among French chronic kidney disease patients: a case-control study. BMC Nephrol. 2020 Feb 26;21(1):63. doi: 10.1186/s12882-020-01722-y. PMID 32101140